CLINICAL TRIAL: NCT05002569
Title: A Phase 3, Randomized, Double-blind Study of Adjuvant Immunotherapy With Nivolumab + Relatlimab Fixed-dose Combination Versus Nivolumab Monotherapy After Complete Resection of Stage III-IV Melanoma
Brief Title: A Study to Assess Adjuvant Immunotherapy With Nivolumab Plus Relatlimab Versus Nivolumab Alone After Complete Resection of Stage III-IV Melanoma
Acronym: RELATIVITY-098
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to meet protocol objectives
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA224-098; 2021-001641-13 (EudraCT Number)
Expanded Access: NCT05170685 (No longer available)
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Melanoma; Relatlimab; Nivolumab; Opdivo
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab Plus Relatlimab (Experimental): Combination
  Interventions: Biological: Nivolumab + Relatlimab Fixed Dose Combination
- Arm B: Nivolumab (Experimental): Monotherapy
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm B: Nivolumab
Biological: Nivolumab + Relatlimab Fixed Dose Combination — Specified dose on specified days
  Other Names: BMS-986213; Opdualag
  Arms: Arm A: Nivolumab Plus Relatlimab

SUMMARY:
The purpose of this study is to assess nivolumab plus relatlimab fixed-dose combination (FDC) versus nivolumab alone in participants with completely resected stage III-IV melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with either Stage IIIA (> 1 mm tumor in lymph node)/B/C/D or Stage IV melanoma by American Joint Committee on Cancer (AJCC) v8 and have histologically confirmed melanoma that is completely surgically resected (free of disease) with negative margins in order to be eligible
* Participants ≥ 18 years of age must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1. Adolescent participants between 12 and < 18 years of age must have a Lansky/Karnofsky performance score ≥ 80%
* Complete resection must be performed within 90 days prior to randomization
* All participants must have disease-free status documented by a complete physical examination within 14 days prior to randomization and imaging studies within 35 days prior to randomization
* Tumor tissue must be provided for biomarker analyses

Exclusion Criteria:

* History of ocular melanoma
* Untreated/unresected CNS metastases or leptomeningeal metastases
* Active, known, or suspected autoimmune disease
* Participants with serious or uncontrolled medical disorder
* Prior immunotherapy treatment for any prior malignancy: No prior immunotherapies are permitted
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 4 weeks prior to screening
* History of myocarditis, regardless of etiology.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1093 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (184):
- United States (43):
  - Local Institution - 0176, Birmingham, Alabama
  - Local Institution - 0164, Springdale, Arkansas
  - Local Institution - 0200, Los Angeles, California
  - Local Institution - 0185, Palo Alto, California
  - Local Institution - 0162, San Francisco, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Local Institution - 0138, Aurora, Colorado
  - Local Institution - 0166, Washington D.C., District of Columbia
  - Local Institution - 0243, Miami, Florida
  - Washington University School Of Medicine, Miami, Florida
  - Local Institution - 0179, Pensacola, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center, Tampa, Florida
  - Local Institution - 0191, Atlanta, Georgia
  - Local Institution - 0148, Atlanta, Georgia
  - Local Institution - 0202, Chicago, Illinois
  - Local Institution - 0177, Peoria, Illinois
  - Local Institution - 0223, Fort Wayne, Indiana
  - University of Iowa-Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Local Institution - 0178, Westwood, Kansas
  - Dana-Farber Cancer Institute-Melanoma, Boston, Massachusetts
  - Local Institution - 0258, Ann Arbor, Michigan
  - Local Institution, Grand Rapids, Michigan
  - Local Institution - 0133, Minneapolis, Minnesota
  - Local Institution - 0139, Hackensack, New Jersey
  - Local Institution - 0206, Morristown, New Jersey
  - Local Institution - 0140, New York, New York
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - Local Institution - 0210, New York, New York
  - Local Institution - 0130, Charlotte, North Carolina
  - Local Institution - 0145, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Local Institution - 0141, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C, Columbus, Ohio
  - Local Institution - 0267, Allentown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0125, Pittsburgh, Pennsylvania
  - Local Institution - 0171, Charleston, South Carolina
  - Local Institution - 0147, Germantown, Tennessee
  - Local Institution - 0183, Nashville, Tennessee
  - Local Institution - 0146, Austin, Texas
  - Local Institution - 0163, Dallas, Texas
  - Local Institution - 0172, Houston, Texas
  - Local Institution - 0137, Fairfax, Virginia
- Argentina (5):
  - Local Institution - 0003, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0005, Buenos Aires, Distrito Federal
  - Local Institution - 0001, CABA, Distrito Federal
  - Local Institution - 0002, Ciudad de Buenos Aires, Distrito Federal
  - Local Institution - 0004, Córdoba
- Australia (12):
  - Local Institution - 0030, Waratah, New South Wales
  - Local Institution - 0252, Westmead, New South Wales
  - Local Institution - 0032, Wollstonecraft, New South Wales
  - Local Institution - 0254, Tiwi, Northern Territory
  - Local Institution - 0028, Brisbane, Queensland
  - Local Institution - 0027, Southport, Queensland
  - Local Institution - 0250, Woodville, South Australia
  - Local Institution - 0035, Ballarat, Victoria
  - Local Institution - 0253, Heidelberg, Victoria
  - Local Institution - 0031, Melbourne, Victoria
  - Local Institution - 0251, Murdoch, Western Australia
  - Local Institution - 0029, Perth, Western Australia
- Austria (3):
  - Local Institution - 0082, Graz, Styria
  - Local Institution - 0086, Salzburg
  - Local Institution - 0084, Vienna
- Belgium (4):
  - Local Institution - 0110, Brussels
  - Local Institution - 0105, Brussels
  - Local Institution - 0109, Liège
  - Local Institution - 0106, Wilrijk
- Brazil (10):
  - Local Institution - 0072, Fortaleza, Ceará
  - Local Institution - 0068, Vitória, Espírito Santo
  - Local Institution - 0071, Salvador, Estado de Bahia
  - Local Institution - 0047, Belo Horizonte, Minas Gerais
  - Local Institution - 0056, Ijuí, Rio Grande do Sul
  - Local Institution - 0257, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0049, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0048, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0070, Barretos, São Paulo
  - Local Institution - 0058, Rio de Janeiro
- Canada (7):
  - Local Institution - 0155, Edmonton, Alberta
  - Local Institution - 0175, Vancouver, British Columbia
  - Local Institution - 0197, Halifax, Nova Scotia
  - Local Institution - 0159, Montreal, Quebec
  - Local Institution - 0158, Montreal, Quebec
  - Local Institution - 0160, Québec, Quebec
  - Local Institution - 0198, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0013, Santiago, Santiago Metropolitan
  - Local Institution - 0006, Santiago, Santiago Metropolitan
  - Local Institution - 0014, Santiago, Santiago Metropolitan
- China (23):
  - Local Institution - 0221, Hefei, Anhui
  - Local Institution - 0259, Beijing, Beijing Municipality
  - Local Institution - 0261, Beijing, Beijing Municipality
  - Local Institution - 0214, Beijing, Beijing Municipality
  - Local Institution - 0241, Chongqing, Chongqing Municipality
  - Local Institution - 0245, Fuzhou, Fujian
  - Local Institution - 0217, Guangzhou, Guangdong
  - Local Institution - 0226, Zhengzhou, Henan
  - Local Institution - 0237, Wuhan, Hubei
  - Local Institution - 0239, Wuhan, Hubei
  - Local Institution - 0234, Changsha Shi, Hunan
  - Local Institution - 0215, Nanjing, Jiangsu
  - Local Institution - 0225, Nanjing, Jiangsu
  - Local Institution - 0224, Nanchang, Jiangxi
  - Local Institution - 0219, Changchun, Jilin
  - Local Institution - 0242, Shenyang, Liaoning
  - Local Institution - 0230, Chengdu, Sichuan
  - Local Institution - 0263, Tianjin, Tianjin Municipality
  - Local Institution - 0228, Ürümqi, Xinjiang
  - Local Institution - 0222, Kunming, Yunnan
  - Local Institution - 0220, Hangzhou, Zhejiang
  - Local Institution - 0216, Hangzhou, Zhejiang
  - Local Institution - 0244, Taiyuan
- Czechia (4):
  - Local Institution - 0156, Brno
  - Local Institution - 0091, Hradec Králové
  - Local Institution - 0026, Ostrava
  - Local Institution - 0062, Prague
- Denmark (4):
  - Local Institution - 0016, Aarhus, Central Jutland
  - Local Institution - 0022, Aalborg
  - Local Institution - 0018, Copenhagen
  - Local Institution - 0020, Odense
- Finland (3):
  - Helsinki University Hospital Adult ICU PPDS, Helsinki
  - Local Institution - 0019, Tampere
  - Local Institution - 0015, Turku
- France (7):
  - Local Institution - 0040, Villejuif, Val-de-Marne
  - Local Institution - 0043, Dijon
  - Local Institution - 0044, Marseille
  - Local Institution - 0039, Nantes
  - Local Institution - 0042, Paris
  - Local Institution - 0041, Pierre-Bénite
  - Local Institution - 0046, Toulouse
- Germany (12):
  - Local Institution - 0092, Tübingen, Baden-Wurttemberg
  - Local Institution - 0079, Hanover, Lower Saxony
  - Local Institution - 0073, Buxtehude
  - Local Institution - 0077, Dresden
  - Local Institution - 0074, Erlangen
  - Local Institution - 0131, Essen
  - Local Institution - 0081, Gera
  - Local Institution - 0075, Heidelberg
  - Local Institution - 0078, Lübeck
  - Local Institution - 0083, Minden
  - Local Institution - 0076, Munich
  - Local Institution - 0080, Würzburg
- Greece (3):
  - Local Institution - 0114, Athens
  - Local Institution - 0113, Neo Faliro
  - Local Institution - 0112, Thessaloniki
- Israel (4):
  - Local Institution - 0199, Petah Tikva, Central District
  - Local Institution - 0118, Jerusalem, Jerusalem
  - Local Institution - 0116, Afula
  - Local Institution - 0117, Ramat Gan
- Italy (7):
  - Local Institution - 0115, Milan
  - Local Institution - 0268, Milan
  - Local Institution - 0123, Milan
  - Local Institution - 0119, Napoli
  - Local Institution - 0120, Padua
  - Local Institution - 0122, Perugia
  - Local Institution - 0121, Siena
- Mexico (4):
  - Local Institution - 0021, Zapopan, Jalisco
  - Local Institution - 0100, Benito Juárez, Mexico City
  - Local Institution - 0093, México, Nuevo León
  - Local Institution - 0098, Oaxaca City
- Norway (3):
  - Local Institution - 0009, Lørenskog, Akershus
  - Local Institution - 0023, Stavanger, Rogaland
  - Local Institution - 0017, Oslo
- Local Institution - 0249, Coimbra, Portugal
- Romania (4):
  - Local Institution - 0170, Brasov
  - Local Institution - 0065, Cluj-Napoca
  - Local Institution - 0066, Craiova
  - Local Institution - 0064, Floresti/ Cluj
- Spain (6):
  - Local Institution - 0188, Badajoz
  - Local Institution - 0201, Barcelona
  - Local Institution - 0151, Donostia / San Sebastian
  - Local Institution - 0153, Granada
  - Local Institution - 0150, Madrid
  - Local Institution - 0152, Valencia
- Sweden (3):
  - Local Institution - 0010, Gothenburg
  - Local Institution - 0011, Lund
  - Local Institution - 0012, Solna
- Switzerland (3):
  - Local Institution - 0085, Basel
  - Local Institution - 0087, Chur
  - Local Institution - 0090, Zurich
- United Kingdom (6):
  - Local Institution - 0101, Nottingham, Nottinghamshire
  - Local Institution - 0102, Bristol
  - Local Institution - 0187, Glasgow
  - Local Institution - 0154, Newcastle upon Tyne
  - Local Institution - 0232, Oxford
  - Local Institution - 0127, Southampton

REFERENCES:
- [Derived] Long GV, Garnett-Benson C, Dolfi S, Ascierto PA, Guo J, Tarhini AA, Chandra S, Munoz-Couselo E, Del Vecchio M, de Melo AC, Callahan M, Gogas H, Dummer R, Schadendorf D, Koelblinger P, Quereux G, Thomas I, Yu JX, Fisher A, Wang B, Djidel P, Chouzy A, Semaan M, Chen B, Cheong AMY, Tawbi HA. Adjuvant nivolumab and relatlimab in stage III/IV melanoma: the randomized phase 3 RELATIVITY-098 trial. Nat Med. 2025 Dec;31(12):4301-4309. doi: 10.1038/s41591-025-04032-8. Epub 2025 Oct 18. PMID 41109920
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1093 participants randomized and 1088 treated.
Groups:
- Treatment 1: nivolumab 480 mg and relatlimab 160 mg IV every 4 weeks (Q4W)
- Treatment 2: nivolumab 480 mg IV Q4W
Period: Randomized
Arm/Group | Treatment 1 | Treatment 2
Started | 547 | 546
Completed (Treated) | 543 | 545
Not Completed | 4 | 1
Not completed — Withdrew Consent | 3 | 0
Not completed — No longer meets study criteria | 0 | 1
Not completed — AE unrelated to study drug | 1 | 0
Period: Treatment Period
Arm/Group | Treatment 1 | Treatment 2
Started | 543 | 545
Completed | 283 | 327
Not Completed | 260 | 218
Not completed — Requested to Discontinue | 26 | 5
Not completed — Withdrew Consent | 7 | 1
Not completed — Study Drug Toxicity | 114 | 64
Not completed — AE unrelated to study drug | 6 | 12
Not completed — Disease Recurrence | 102 | 128
Not completed — Other Reasons | 4 | 7
Not completed — Death | 1 | 1
Period: Follow Up
Arm/Group | Treatment 1 | Treatment 2
Started | 543 | 545
Completed | 1 | 5
Not Completed | 542 | 540
Not completed — Death | 78 | 69
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrew consent | 17 | 16
Not completed — Other Reasons | 444 | 452

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 547 | 546 | 1093
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (14.16) | 57.6 (13.34) | 57.4 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 231 | 451
  Male | 327 | 315 | 642
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 39 | 85
  Not Hispanic or Latino | 280 | 269 | 549
  Unknown or Not Reported | 221 | 238 | 459
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 37 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 491 | 497 | 988
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS)
Description: RFS is defined as the time between the date of randomization and the first date of documented recurrence (local, regional, distant, new primary melanoma) or death due to any cause, whichever occurs first.
Time Frame: Approximately 27.5 Months
Population: All Randomized Participants
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 547 | 546
Months | NA [0 to 37.7] — Insufficient number of participants with events to calculate via KM Methodology | 33.84 [0 to 37.7]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Approximately 27.5 Months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 547 | 546
Months | NA [NA to NA] — Insufficient number of participants with events to calculate via KM Methodology | NA [NA to NA] — Insufficient number of participants with events to calculate via KM Methodology

3. Secondary Outcome: Distant Metastasis Free Survival (DMFS)
Description: DMFS is defined as the time between the date of randomization and the date of first distant metastasis or date of death due to any cause, whichever occurs first.
Time Frame: Approximately 27.5 Months
Population: All Randomized Participants with Resected Stage 3/4a/4b Melanoma at study entry
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 499 | 494
Months | NA [NA to NA] — Insufficient number of participants with events to calculate via KM Methodology | NA [33.84 to NA] — Insufficient number of participants with events to calculate via KM Methodology

4. Secondary Outcome: Progression Free Survival on Next-Line Systemic Therapy (PFS2)
Description: PFS2 defined as time from randomization to second recurrence/objective disease progression on next-line systemic therapy per investigator, or death from any cause, whichever occurs first.
Time Frame: Approximately 27.5 Months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 547 | 546
Months | NA [NA to NA] — Insufficient number of participants with events to calculate via KM Methodology | NA [NA to NA] — Insufficient number of participants with events to calculate via KM Methodology

5. Secondary Outcome: Number of Participants With Safety Related Events
Description: Safety related events encompass the following measures: Adverse events (AEs), Serious AEs, AEs leading to discontinuation, Drug-Related AEs and Deaths.
  An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
  An SAE is an AE which:
  * Results in death
  * Is life threatening
  * Requires hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Time Frame: Approximately 27.5 Months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 543 | 545
Participants
  AEs | 522 | 520
  Drug-Related AEs | 483 | 438
  Serious AEs | 132 | 78
  AEs leading to discontinuation | 102 | 65
  Deaths | 83 | 76

6. Secondary Outcome: Number of Participants With Select AEs
Description: Select AEs will be reported as AEs per organ class.
  Organ classes which will be reported:
  * Gastrointestinal
  * Hepatic
  * Pulmonary
  * Renal
  * Skin
  * Hypersensitivity/Infusion reaction
Time Frame: Approximately 27.5 Months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 543 | 545
Participants
  Gastrointestinal | 115 | 120
  Hepatic | 108 | 86
  Pulmonary | 11 | 13
  Renal | 33 | 21
  Skin | 244 | 240
  Hypersensitivity/Infusion Reaction | 37 | 26

7. Secondary Outcome: Number of Participants With Endocrine Related Immune Mediated AEs
Description: Immune-mediated adverse events are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity.
Time Frame: Approximately 27.5 Months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 543 | 545
Participants
  Adrenal Insufficiency | 33 | 9
  Hypothyroidism/Thyroiditis | 158 | 93
  Hypothyroidism | 152 | 82
  Thyroiditis | 18 | 14
  Diabetes Melitus | 11 | 8
  Hyperthyroidism | 96 | 56
  Hypophysitis | 51 | 13

8. Secondary Outcome: Number of Participants With Non-endocrine Related Immune Mediated AEs
Description: as for outcome 7
Time Frame: Approximately 27.5 Months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 543 | 545
Participants
  Pneumonitis | 8 | 10
  Diarrhea/colitis | 28 | 21
  Hepatitis | 26 | 17
  Nephritis and Renal Dysfunction | 3 | 3
  Rash | 49 | 40
  Hypersensitivity | 12 | 2

9. Secondary Outcome: Laboratory Abnormalities for Specific Thyroid Tests
Description: Number of participants with laboratory abnormalities in specific thyroid tests.
Time Frame: Approximately 27.5 Months
Population: All Treated Participants with at least one on treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 524 | 534
Participants
  TSH > ULN | 229 | 159
  TSH > ULN WITH TSH ≤ ULN AT BASELINE | 193 | 124
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 148 | 74
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES ≥ LLN | 168 | 124
  TSH > ULN WITH FT3/FT4 TEST MISSING | 52 | 28
  TSH < LLN | 198 | 131
  TSH <LLN WITH TSH ≥ LLN AT BASELINE | 180 | 123
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 119 | 72
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES ≤ ULN | 117 | 85
  TSH < LLN WITH FT3/FT4 TEST MISSING | 27 | 19

ADVERSE EVENTS:
Time Frame: Adverse Events, Serious Adverse Events and All-Cause mortality: Approximately 27.5 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 86/547 | 76/546
Serious Adverse Events (participants affected / at risk) | 174/543 | 121/545
Other Adverse Events (participants affected / at risk) | 489/543 | 473/545
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=543) | Treatment 2 (N=545)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Sarcoidosis of lymph node (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Autoimmune myocarditis (Cardiac disorders) | 3 | 3
Cardiac failure (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocarditis (Cardiac disorders) | 8 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hypophysitis (Endocrine disorders) | 13 | 2
Hypopituitarism (Endocrine disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 1 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 2 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1
Amaurosis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Eosinophilic gastritis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 4 | 3
Immune-mediated gastritis (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 2
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Immune-mediated polyserositis (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Serositis (General disorders) | 1 | 0
Sudden death (General disorders) | 2 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 4 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 2
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 2
Campylobacter colitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Complicated appendicitis (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Kidney infection (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication circulatory (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 2 | 0
Norovirus test positive (Investigations) | 0 | 1
Troponin I increased (Investigations) | 1 | 1
Troponin T increased (Investigations) | 2 | 1
Troponin increased (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 6 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 9 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 12
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Immune-mediated myasthenia gravis (Nervous system disorders) | 0 | 1
Immune-mediated myelitis (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 4 | 0
Myelitis transverse (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Sarcoid-like reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin cosmetic procedure (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=543) | Treatment 2 (N=545)
Anaemia (Blood and lymphatic system disorders) | 36 | 25
Hyperthyroidism (Endocrine disorders) | 96 | 60
Hypophysitis (Endocrine disorders) | 37 | 10
Hypothyroidism (Endocrine disorders) | 150 | 85
Abdominal pain (Gastrointestinal disorders) | 31 | 24
Constipation (Gastrointestinal disorders) | 44 | 32
Diarrhoea (Gastrointestinal disorders) | 114 | 117
Dry mouth (Gastrointestinal disorders) | 59 | 36
Nausea (Gastrointestinal disorders) | 86 | 54
Vomiting (Gastrointestinal disorders) | 29 | 31
Asthenia (General disorders) | 68 | 69
Fatigue (General disorders) | 161 | 161
Oedema peripheral (General disorders) | 30 | 23
Pyrexia (General disorders) | 39 | 32
COVID-19 (Infections and infestations) | 78 | 110
Nasopharyngitis (Infections and infestations) | 31 | 32
Infusion related reaction (Injury, poisoning and procedural complications) | 29 | 19
Alanine aminotransferase increased (Investigations) | 69 | 57
Aspartate aminotransferase increased (Investigations) | 59 | 49
Blood creatine phosphokinase increased (Investigations) | 27 | 35
Decreased appetite (Metabolism and nutrition disorders) | 46 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 29 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 100 | 110
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 47
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 30
Dizziness (Nervous system disorders) | 29 | 29
Headache (Nervous system disorders) | 74 | 94
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 59
Pruritus (Skin and subcutaneous tissue disorders) | 112 | 116
Rash (Skin and subcutaneous tissue disorders) | 99 | 86
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 | 20
Hypertension (Vascular disorders) | 26 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT05002569/Prot_SAP_000.pdf